CLINICAL TRIAL: NCT05424133
Title: Comparative Effects of Active Cycle of Breathing Technique and High Frequency Chest Wall Oscillation in Chronic Obstructive Pulmonary Disease Patients
Brief Title: ACBT and High Frequency Chest Wall Oscillations in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0321
Record Dates: First submitted 2022-05-23; First posted 2022-06-21 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chest wall oscillation; Respiration; Pulmonary disease; Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration; Lung Diseases | interventions — Chest Wall Oscillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cycle of breathing technique (Experimental): Group A will receive Active cycle of breathing technique with routine chest physiotherapy.
  Interventions: Other: Active cycle of breathing
- High frequency chest wall oscillation (Active Comparator): Group B will receive High frequency chest wall oscillations with routine chest physiotherapy
  Interventions: Other: High frequency chest wall oscillation

INTERVENTIONS:
Other: High frequency chest wall oscillation — High frequency chest wall oscillations at 13-15Hz oscillating frequency for 20 minutes twice a day for 4 weeks.
  Arms: High frequency chest wall oscillation
Other: Active cycle of breathing — Active cycle of breathing technique and it will performed twice a day for 4 week intervention period for 20 minutes
  Arms: Active cycle of breathing technique

SUMMARY:
Chronic obstructive pulmonary disease (COPD) patients with mucus hyper secretion tend to demonstrate increased frequency of infective exacerbations and a steeper slope of decline in lung function. Enhanced mucosal clearance with high frequency chest wall oscillation (HFCWO) devices previously used in cystic fibrosis and bronchiectasis patients may offer the opportunity for community based, self-managed therapy to improve quality of life and lung function. The aim of this study is to compare effects of active cycle of breathing and high frequency chest wall oscillations in chronic obstructive pulmonary disease .This study will be a Randomized Clinical trial and will be conducted at Physical Therapy Department of DHQ Hospital NAROWAL. The study will be completed within the time duration of six months. Consecutive sampling technique will be used to collect the data. A sample size of Total 42 patients will be taken in this study. Patients will be divided into two groups. BODE Index will be used as outcome measurement tool. Group A will receive the Active cycle of breathing technique and it will performed twice a day for 4 week intervention period for 20 minutes. Group B will receive high frequency chest wall oscillations at 13-15Hz oscillating frequency for 20 minutes twice a day for 4 weeks. The collected data will be analyzed on SPSS - 25.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clear consciousness ,stable vital sign, and ability to cooperate
* Stage 3-4 COPD according to GOLD criteria
* Adult patients
* Patient who had given informed consent

Exclusion Criteria:

* Need for invasive mechanical ventilation
* Active lung tuberculosis
* Chest wall trauma
* Thoracic or abdominal operations in last three months.
* Presence of cardiac pacemaker, artificial stunt or heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
BODE Index | 4th week
  The BODE index is a tool that is used by healthcare professionals to predict the mortality rate from chronic obstructive pulmonary disease (COPD) The final score of the BODE index ranges from 0 to 10 points; higher the index value, the worse is the patient's condition. The participants were divided into four quartiles for the analysis according to their BODE index score, Quartile I is a score of 0-2 points, quartile II 3-4 points, quartile III v 5-6 points, and quartile IV is a score of 7-10 points.
  BODE Index Scale score at baseline and 4th week

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital Narowal, Narowal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen M, Li Y, Ding X, Xu L, Li F, Lin H. Effect of active cycle of breathing techniques in patients with chronic obstructive pulmonary disease: a systematic review of intervention. Eur J Phys Rehabil Med. 2020 Oct;56(5):625-632. doi: 10.23736/S1973-9087.20.06144-4. Epub 2020 May 13. PMID 32397703
- [Background] Barto TL, Maselli DJ, Daignault S, Stiglich J, Porter J, Kraemer C, Hansen G. Real-life experience with high-frequency chest wall oscillation vest therapy in adults with non-cystic fibrosis bronchiectasis. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620932508. doi: 10.1177/1753466620932508. PMID 32538317
- [Background] Ntritsos G, Franek J, Belbasis L, Christou MA, Markozannes G, Altman P, Fogel R, Sayre T, Ntzani EE, Evangelou E. Gender-specific estimates of COPD prevalence: a systematic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2018 May 10;13:1507-1514. doi: 10.2147/COPD.S146390. eCollection 2018. PMID 29785100
- [Background] Weycker D, Hansen GL, Seifer FD. Outcomes with high-frequency chest wall oscillation among patients with non-CF bronchiectasis or COPD. American Thoracic Society. 2017. 7. Sievert CE, Beaner BCA, Sievert C. Using High Frequency Chest Wall Oscillation in a Bronchiectasis Patient Population: An Outcomes-Based Case Review. Respiratory Therapy. 2016;10:01.
- [Background] Allam NM, Badawy MM. Does High-Frequency Chest Wall Oscillation Have an Impact on Improving Pulmonary Function in Patients With Smoke Inhalation Injury? J Burn Care Res. 2021 Mar 4;42(2):300-304. doi: 10.1093/jbcr/iraa147. PMID 32860696
- [Background] Gonzalez-Bellido V, Velaz-Baza V, Blanco-Moncada E, Del Carmen Jimeno Esteo M, Cuenca-Zaldivar JN, Colombo-Marro A, Donadio MVF, Torres-Castro R. Immediate Effects and Safety of High-Frequency Chest Wall Compression Compared to Airway Clearance Techniques in Non-Hospitalized Infants With Acute Viral Bronchiolitis. Respir Care. 2021 Mar;66(3):425-433. doi: 10.4187/respcare.08177. Epub 2020 Nov 3. PMID 33144386
- [Background] Shen MD, Guo LR, Li YW, Gao RT, Sui X, Du Z, Xu LQ, Shi HY, Ni YY, Zhang X, Pang Y, Zhang W, Yu TZ, Li F. Role of the active cycle of breathing technique combined with phonophoresis for the treatment of patients with chronic obstructive pulmonary disease (COPD): study protocol for a preliminary randomized controlled trial. Trials. 2021 Mar 23;22(1):228. doi: 10.1186/s13063-021-05184-x. PMID 33757568